CLINICAL TRIAL: NCT06933875
Title: Promoting Palliative Care for People With Heart Failure: The P3HF Pilot Study
Brief Title: Promoting Palliative Care for People With Heart Failure
Acronym: P3HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000038269; 1R34HL174885-01 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Palliative Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Providers who care for people hospitalized with heart failure at the two study sites will be recruited. Providers will be selected via retrospective chart review by study investigators. Eligibility of patients will be assessed automatically by an existing Epic build and will not involve any human intervention. When a provider opens the order entry screen of the patient's medical record, this build will examine the record for all inclusion and exclusion criteria. Those who meet criteria will be automatically enrolled and placed into a randomization group based on the randomization status of their current provider at the time of enrollment. Target sample size is 70 providers, 700-1400 participants and 15 Level 2 providers (providers potentially impacted by the tool).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical Decision Support (CDS) Tool (Experimental): Providers will use the CDS tool to deliver prognostic information and evidence-based decision support at the point of care for timely referral to palliative care for participants hospitalized with heart failure.
  Interventions: Behavioral: Clinical Decision Support Tool
- Standard of Care (No Intervention): Providers will provide usual standard of care for participants hospitalized with heart failure.
- Level 2 providers (Experimental): Level 2 providers are providers potentially impacted by the tool. Level 2 providers will participate in one interview.
  Interventions: Behavioral: Clinical Decision Support Tool

INTERVENTIONS:
Behavioral: Clinical Decision Support Tool — Deliver prognostic information and evidence-based decision support at the point of care
  Arms: Clinical Decision Support (CDS) Tool; Level 2 providers

SUMMARY:
This project will develop and test a novel clinical decision support tool (CDS) that encourages timely referral to palliative care for people hospitalized with heart failure. This intervention will incorporate an existing, validated 1-year mortality risk model into a CDS to deliver prognostic information and evidence-based decision support at the point of care. Thus, this research may lead to improved care-concordant and goal-directed care for people with heart failure.

DETAILED DESCRIPTION:
Healthcare providers will encounter the tool during the routine care of their hospitalized patients. Providers randomized to the intervention arm will receive training on the use of the tool and complete one post-trial survey. Providers randomized to the intervention arm will also have the opportunity to participate in 1 post-trial interview. Level 2 providers will participate in one interview.

ELIGIBILITY:
Inclusion Criteria:

Healthcare providers must meet the following criteria:

* Are an attending physician, fellow, or resident, advanced practice nurse, or physician associate
* Has ordering privileges
* Are members of one of the hospitals' admitting teams (e.g., hospitalist service, cardiology service)
* Anticipate employment at one of the two study sites for the 15-month trial period.

Or

* Palliative care team member
* Hospital administrator/quality and safety personnel

Patients of providers enrolled in the study must meet the following criteria for heart failure during hospitalization:

* N-terminal pro-B-type natriuretic peptide values of >500 pg/ml
* Not pregnant at the time of admission.
* Received intravenous diuretics within 24 hours of admission.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1485 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean System Usability Scale score | up to 15 months
  System Usability Scale, 10-item Likert questionnaire. Total score range 0-100. Higher values indicate higher usability
Mean Acceptability of Intervention Measure score | up to 15 months
  Acceptability of Intervention Measure, 4-item questionnaire. Total score range 1-4. Higher values indicate higher acceptability.
Mean Appropriateness of Intervention Measure score | up to 15 months
  Appropriateness of Intervention Measure, 4-item questionnaire. Total score range 1-4. Higher values indicate higher appropriateness.
Mean Feasibility of Intervention Measure score | up to 15 months
  Feasibility of Intervention Measure, 4-item questionnaire. Total score range 1-4. Higher values indicate higher feasibility.

SECONDARY OUTCOMES:
Referral to Specialist Palliative Care | up to 15 months
  Proportion of participants who are referred to Specialist Palliative Care
Consultation by Specialist Palliative Care | up to 15 months
  Proportion of participants who have a completed consultation order by Specialist Palliative Care
Advance Care Plan Documentation | up to 15 months
  Proportion of participants who have a documented Advance Care Plan
Participants enrolled in hospice | up to 15 months
  Proportion of participants enrolled in hospice during hospitalization
Mean hospital length of stay | up to 15 months
  Mean hospital length of stay in days
Participants readmitted to hospital | up to 15 months
  Proportion of participants with 30-day hospital readmission

CONTACTS AND LOCATIONS:
Overall Officials: Shelli Feder, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital Saint Raphael, New Haven, Connecticut
  - Yale New Haven Hospital York Street, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No